CLINICAL TRIAL: NCT04430907
Title: Increasing Human Papillomavirus Vaccination in Postpartum Women at Penn State Hershey Medical Center
Brief Title: HPV Vaccine in Postpartum Women
Status: Withdrawn | Type: Observational
Why Stopped: Revising protocol.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stacey Milunic, Associate Professor, Family and Community Medicine, Milton S. Hershey Medical Center
Other Study IDs: 13831
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: HPV Infection
Keywords: HPV vaccination; cervical cancer; postpartum
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Vaccine Accepting: This group will receive the HPV vaccine in the inpatient postpartum period prior to discharge from the hospital.
  Interventions: Biological: HPV 9-valent Vaccine, Recombinant
- Vaccine Rejecting: This group will not receive the HPV vaccine in the inpatient postpartum period prior to discharge from the hospital.

INTERVENTIONS:
Biological: HPV 9-valent Vaccine, Recombinant — After consent, participants will complete an intake survey confirming eligibility. Participants will also complete a survey asking about knowledge, attitudes, and beliefs around vaccination, including HPV vaccination, as well as breastfeeding intentions.
  After survey completion, the participant will be asked if they would like to be administered the HPV vaccine, Gardasil 9. If participants do not agree, they will be contacted 1-week later for the follow-up survey. If participants do agree, the project coordinator will notify the study physician, who will place an order for the vaccine. The vaccine will be administered to the patient prior to discharge from the hospital. Participants will be contacted 1-week later for the follow-up survey.
  Other Names: Gardasil-9
  Groups: Vaccine Accepting

SUMMARY:
The purpose of this study is to determine the acceptability of HPV vaccination in postpartum women in Central Pennsylvania. Participants will be recruited while inpatient in the postpartum unit. Participants will complete a survey asking about knowledge, attitudes, and beliefs around vaccination, including HPV vaccination, as well as breastfeeding intentions. After survey completion, the participant will have the option to receive the HPV vaccine, Gardasil 9, prior to discharge from the hospital. All participants will then be contacted 1- week later for the follow-up survey.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if postpartum women serve as a potential population to target in order to increase human papillomavirus (HPV) vaccination in Central Pennsylvania.

Despite being available for almost a decade, uptake of the HPV vaccine in the US remains below other countries, including England, Scotland, and Australia. In fact, in 2017, only 67% of US girls aged 13-17 had obtained even one dose of the HPV vaccine series. Due to low rates of HPV vaccination in the United States and Central Pennsylvania, effective interventions are needed to help increase these rates.

While vaccination is recommended at a younger age, it is effective among women 18-25 years old. Based on clinical trial data, giving the vaccine to this age group has resulted in reduced abnormal Pap test findings, referral for colposcopy, and treatment related to abnormal cervical cytology. However, the HPV vaccine is not usually discussed during prenatal care or routinely administered during pregnancy. Previous studies have shown that offering other vaccines postpartum (e.g. tetanus or pertussis) has been successful.

By offering the vaccine to this demographic group, the investigators could potentially discover an untapped target population to help increase rates of HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Women postpartum with a live birth at Penn State Hershey Medical Center (PSHMC), either vaginal or cesarean delivery.
2. Women aged 18-26 (inclusive) years
3. Women who are on a Floor Status level of care.
4. Women who have completed 0 or 1 doses of the HPV vaccine STUDY00013831 Approval: 5/8/2020 Page 6 of 24 (V.01/21/2019)
5. Fluent in written and spoken English and other languages in which the Human Subjects Protection Office (HSPO) Consent Short From is available (French, Italian, Russian, Spanish, Vietnamese, Hindi, Chinese and Nepali)

Exclusion Criteria:

1. Women who have completed 2 or 3 doses of the HPV vaccine
2. Hypersensitivity, including severe allergic reactions to yeast (a vaccine component), or after a previous dose of GARDASIL 9 or GARDASIL®.
3. Allergic reaction to amorphous aluminum hydroxyphosphate sulfate or polysorbate 80
4. Women being actively treated for cancer.
5. Have a fever over 100.4 degrees Fahrenheit (38.0 degrees Celsius)
6. Women who are at an ICU level of Care
7. Women who are on a Labor and Delivery Level of Care
8. Women receiving continuous IV magnesium.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women postpartum with a live birth at Penn State Hershey Medical Center (PSHMC), either vaginal or cesarean delivery between the ages of 18-26 (inclusive).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of postpartum women who agree to HPV vaccination | Day 1
  Percentage of women who accept HPV vaccination when offered in the inpatient postpartum setting
Perception of HPV vaccination | Day 8
  Perception of HPV vaccination as measured via Likert scale questions in pre- and post survey. The investigators use a 5-point Likert scale, where '1' means 'strongly disagree', '2' means somewhat disagree, '3' means neither agree or disagree, '4' means somewhat agree, and '5' means 'strongly agree'. The higher the score, the more favorable the outcome.
Satisfaction to receive the HPV vaccine | Day 8
  Patient satisfaction with her decision to receive (or not receive) the HPV vaccine as measured via Likert scale questions in pre and post survey. The investigators use a 5-point Likert scale, where '1' means 'strongly disagree', '2' means somewhat disagree, '3' means neither agree or disagree, '4' means somewhat agree, and '5' means 'strongly agree'. The higher the score, the more favorable the outcome.

SECONDARY OUTCOMES:
Perception of vaccines in general | Day 1
  Perception of vaccines overall (not specific to HPV) as measured via Likert scale questions in pre-survey. The investigators use a 5-point Likert scale, where '1' means 'strongly disagree', '2' means somewhat disagree, '3' means neither agree or disagree, '4' means somewhat agree, and '5' means 'strongly agree'. The higher the score, the more favorable the outcome.
Breastfeeding intentions and practices | Days 1 and 8
  Differences in breastfeeding intentions/practices for women who get HPV vaccine in the postpartum setting versus women who refuse HPV vaccine in the postpartum setting as measured by pre- and post-surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Milunic, MD, Principal Investigator — Penn State College of Medicine

IPD SHARING:
Plan to Share IPD: No